CLINICAL TRIAL: NCT02134626
Title: Simvastatin Effect in Portal Hypertension Measured by Portal Hemodynamic Gradient and Azygos Vein Doppler in Echoendoscopy
Brief Title: Simvastatin Effect on Portal Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Guilherme Rezende, Associate Professor of the Medical Faculty, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: simvhp01
Record Dates: First submitted 2014-04-04; First posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Portal Hypertension; Esophageal Varices; Liver Cirrhosis
Keywords: Portal Hypertension; Hepatic Venous Pressure Gradient; Esophageal Varices; Liver Cirrhosis; Simvastatin; Nitric oxide; HVPG
MeSH Terms: conditions — Hypertension, Portal; Esophageal and Gastric Varices; Liver Cirrhosis | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin (Experimental): Arm 1: Simvastatin 40mg / pill, one pill once a day for three months
  Interventions: Drug: Simvastatin
- Placebo pill (Placebo Comparator): Arm 2: Placebo one pill once a day for three months
  Interventions: Drug: Placebo pill

INTERVENTIONS:
Drug: Simvastatin — 40mg / pill, one pill orally once a day for three months
  Arms: Simvastatin
Drug: Placebo pill
  Arms: Placebo pill

SUMMARY:
It´s a clinical research of the effects in portal hypertension caused by simvastatin. We are going to use the hepatic venous pressure gradient(HVPG) measurement and the azygos flow at echoendoscopy to evaluate the benefits of the drug. Preliminary studies demonstrated that simvastatin can lower portal pressure.

DETAILED DESCRIPTION:
The simvastatin can target the liver enhancing nitric oxide intra-hepatic and lowering resistance that may be responsible for most of cirrhosis complications. Indeed, the potential use of this drug may ameliorate the HVPG and azygos flow. Portal hypertension is responsible for most of the cases of death in cirrhosis. The esophageal varices, ascites and hepatorenal syndrome are the most harmful consequences of cirrhosis that should be prevented. In that way, simvastatin appears as a promising therapy.The study will include two groups of patients using aleatory randomization and one group will receive simvastatin while the other will receive placebo blindly. At the start and at the end of the study the patients will be submitted to HVPG measurement and azygous vein flow measure.

The endpoints will be the normalization of HVPG or lower significantly(20% or more.

The patients will be followed for 6 months after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Portal hypertension: esophageal varices, ascites, splenomegaly or hepatorenal syndrome.

Exclusion Criteria:

* Child-Pugh C decompensated or encephalopathy
* Malignancy except basocellular cancer
* Hepatocarcinoma
* Anti-viral therapy
* HIV
* Prevention of digestive hemorrhage with band ligation or sclerotherapy for the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Hepatic venous pressure gradient (HVPG) in mmHg units | 3 months
  Positive results consist of reduction of the HVPG to values equal or less than 12 mmHg or 20% lower than the first measure

CONTACTS AND LOCATIONS:
Overall Officials: Priscila Pollo-Flores, MD, Master, Principal Investigator — Federal University of Rio de Janeiro - UFRJ
Locations (1):
- Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil